CLINICAL TRIAL: NCT06797726
Title: Feasibility and Efficacy of Cognitive-Behavioral Therapy for Patients With ADHD/Behavioral Addiction Comorbidity: a Pilot Randomized Controlled Trial (ADHDDICT)
Brief Title: Feasibility and Efficacy of Cognitive-Behavioral Therapy for Patients With ADHD/Behavioral Addiction Comorbidity
Acronym: ADHDDICT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Nantes University Hospital (Other); University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR240076
Record Dates: First submitted 2024-11-26; First posted 2025-01-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: ADHD; Behavioral Addiction
Keywords: CBT; Cognitive behavioral therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT group (Experimental): 10 sessions of Cognitive Behavioral Therapy (CBT) Behavioral and Cognitive Therapy (CBT) adapted to comorbidity ADHD/behavioral addiction in remote format (teleconsultation) + routine care (care provided according to the protocols of each center).
  Interventions: Behavioral: Cognitive behavioral therapy
- Control group (No Intervention): routine care (care performed according to protocols of each center)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Session 1: Functional analysis, motivational approach and psycho-education (advantages/disadvantages of consumption ; effect of addiction on mental disorders and interaction ADHD/behavioral addiction) Session 2: Follow-up to psycho-education session 1, treatment plan Session 3: ADHD: compensation strategies; reducing distractibility distractibility Session 4: ADHD: calendar and organization worksheet Session 5: ADHD: mood disorders and emotions Session 6: Recognizing and managing emotions Session 7: Analysis of functional elements in addictive disorder addictive disorders in patients with ADHD Session 8: Risk situations, psycho-education (emotions) Session 9: Managing craving; analysis of the functional elements of of addiction Session 10: Relapse and relapse prevention, problem solving and social pressure
  Arms: CBT group

SUMMARY:
The main objective of this pilot study is to assess preliminary data on the feasibility of CBT and its evaluation in a randomised trial in patients with co-occurring ADHD and behavioural addiction: Evaluation and comparison of the 12-week retention rate of patients randomised to CBT compared with patients in the 'treatment as usual' control arm.

In order to meet the objective, the patient will take part in a standardized assessment, followed by a therapeutic intervention and a new standardized assessment after the intervention. The standardized assessment consists as follows :

* firstly, 7 self-questionnaires to be completed by the patient, lasting around 45 min, aimed at assessing his or her socio-demographic data; current symptoms, quality of life and functional impact related to ADHD; impulsivity, emotion regulation and assessment of possible anxiety-depressive disorders.
* Then the patient will follow the 10 session of cognitivo behavioural psychotherapy.
* At 12-weeks post-inclusion, an assessment visit is carried out during which a battery of tests will be administered. This is followed by a research interview with a professional, aimed at gathering his or her experiences.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 (age ≥ 18 years)
* Patient treated in an outpatient addictology department at the CHU of Brest, Nantes or Tours and presenting an ADHD/behavioral addiction comorbidity
* Patient affiliated to a social security scheme
* For patients treated with methylphenidate: no change in treatment dosage during the previous three months.
* For patients not treated with methylphenidate: no introduction of methylphenidate within the next three months.

Exclusion Criteria:

* Patients with psychotic disorders (assessed by clinician)
* Pregnant or breast-feeding women
* Patients under protective supervision (guardianship or curatorship)
* Persons under court protection
* Persons deprived of their liberty
* Patients who do not meet the eligibility criteria for CBT (e.g., cognitive impairment, hearing impairment).
* Physical inability to participate in CBT sessions (e.g., lack of telephone, foreseeable unavailability).
* Difficulty understanding self-questionnaires, including illiteracy.
* Participation in another interventional research protocol involving another psychotherapeutic or pharmacological intervention that may have an impact on clinical outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Retention rate | At the 12-week
  Proportion of randomized present at the 12-week visit
Adhesion | Between baseline and 12 weeks
  Number of sessions performed between baseline and 12 weeks,
Adhesion | between baseline and 12 weeks
  percentage of patients who attended at least 70% of sessions

SECONDARY OUTCOMES:
Quantitative evaluation of acceptance percentage | At 14 weeks
  Number of randomized patients / number of eligible patients eligible patients
Satisfaction of participants in the Cognitive-behavioural therapy group | At 14 weeks
  only assessed in Cognitive-behavioural therapy group, assessed during an interview with a psychologist (qualitative evaluation)
Perceived benefits | At 14 weeks
  only assessed in Cognitive-behavioural therapy group, assessed during an interview with a psychologist
Collection of difficulties during the therapy | At 14 weeks
  only assessed in Cognitive-behavioural therapy group, assessed during an interview with a psychologist
Assessment of barriers and levers to psychotherapy and cognitive behavioral disorder therapy | At 14 weeks
  Evaluated only for the control group, assessed during an interview with a psychologist
Assessment of patients' perceived needs in terms of psychotherapy | At 14 weeks
  Evaluated only for the control group, assessed during an interview with a psychologist
ADHD symptoms | From baseline up to 12 weeks
  Evaluation will be based on the ASRS-18 (Adult Self-Report Scale) total score. This self-administered questionnaire comprises eighteen questions, six of which are considered to be the most representative of the symptoms associated with ADHD. These six questions, in Part A of the questionnaire, form the core of the ASRS v1.1 screening. Part B contains the remaining twelve questions. The impact of symptoms on different areas of the patient's life is also assessed. Screening is positive when the patient presents at least 4 symptoms with a significant impact among the first 6 items . Each item is rated from 0 to 4, giving a total ASRS-18 score ranging from 0 to 72, with sub-scores for inattention (0 to 36), motor hyperactivity/impulsivity (0 to 20) and verbal hyperactivity/impulsivity (0 to 16).
Quality of life specific to attention-deficit disorder (ADHD) | From baseline up to 12 weeks
  The Adult ADHD Quality of Life scale (AAQOL) will be used during the assessment phases. This tool has good psychometric qualities and assesses four dimensions of quality of life: productivity in daily life, psychological health, relationships and outlook on life. The AAQOL provides a total quality of life score, as well as 4 sub-scores for each dimension. The total score is between 0 and 100, the sub-dimension scores between 0 and 100 (transformed from responses to each of the responses to each of the 29 items ranging from 1 to 5). The higher the score (total and sub-score), the higher, the better the quality of life
Functional impact of attention deficit hyperactivity disorder (ADHD) | From baseline up to 12 weeks
  The Weiss Functional Impairment Rating Scale-Self-Report (WFIRS-S) will be used during the assessment phases. This tool, with good psychometric qualities, assesses the impacts of ADHD in seven domains: family, work life, school life, life skills, self-image, social life and risk-taking. Any item rated "2" or "3" is two standard deviations outside the clinical norms for ADHD and is considered impaired. A conservative threshold for defining impairment in any domain is either two items scored '2', or one item scored '3'. The average item score for most domains is '1', with the exception of 'at-risk activities', which is '0.5'. The average score for each of the 7 dimensions is between 0 and 3.
Craving | From baseline up to 12 weeks
  A visual analog scale (VAS) to assess craving will be used. In the absence of a validated tool to measure craving in a homogeneous way in behavioral addictions, we will ask participants to rate the intensity of craving on a scale from 0 to 10 (0 corresponding to no craving and 10 to maximum craving) and to evaluate the frequency of craving as well as its duration. This type of craving measurement is frequently used in the literature and in addiction research protocols.
Impulsivity | From baseline up to 12 weeks
  The Impulsive Behavior Scale (UPPS-P) will be used during the assessment phases to measure impulsivity. This tool has good psychometric qualities and measures the following sub-dimensions of impulsivity: positive urgency, negative urgency, lack of premeditation, lack of perseverance and sensation seeking. The score for each dimension ranges from 4 to 16; there is no total score. The higher the score (subscales), the higher the impulsivity.
Emotional dysregulation | From baseline up to 12 weeks
  The Difficulties in Emotion Regulation Scale (DERS 36) will be used (during the assessment phases) to evaluate emotional dysregulation. With good psychometric qualities, this scale measures 6 dimensions: unacceptance of negative emotions, difficulty engaging in goal-directed behaviors in the presence of negative emotions, difficulty controlling impulsive behaviors in the presence of negative emotions, restricted access to emotion regulation strategies perceived as effective, emotional awareness and lack of understanding of one's emotions, defined as a lack of emotional clarity. The total score ranges from 36 to 180, with sub-dimensions scores ranging from 6 to 30. The higher the score (total scale and subscales), the greater the emotional dysregulation.
Anxiety symptoms | From baseline up to 12 weeks
  The Hospital Anxiety and Depression scale (HAD) will be used to assess the presence of anxiety and depressive symptoms in participants. This is a variable we wish to control for, in order to verify that anxiety and depressive symptoms are not potential confounding factors in the assessment results. This scale has good psychometric qualities and can be used to assess two dimensions: anxiety symptoms and depressive symptoms. The total score ranges from 0 to 21 for each dimension. For each dimension, the following interpretation can be proposed:
  - 7 or less: no symptoms - 8 to 10: moderate score - 11 to 14: average score 15 to 21: severe score. In practice, a threshold score ≥ 11 for each subscale is retained for a significant anxiety or depression score.
Evolution of psychiatric disorders | At 12 weeks
  Evaluation will be based on MINI-S interview (mini international neuropsychiatric interview, simplified )
Severity of addictive disorders | At 12 weeks
  Evaluation will be based on Clinical Global Impression. The CGI includes two complementary single-item measures that assess the following:
  (a) severity of psychopathology on a scale of 1 to 7 and (b) change from baseline on a similar treatment on a similar seven-point scale. Following a assessment, the CGI can be completed in less than a minute by an experienced experienced assessor. The CGI is used to gather clinical impressions and track clinical clinical progress over time

CONTACTS AND LOCATIONS:
Overall Officials: Servane BARRAULT, Dr, Principal Investigator — CHRU de Tours; Clémence CABLEGUEN, Dr, Principal Investigator — Nantes University Hospital; Morgane GUILLOU, Dr, Principal Investigator — CHU Brest
Locations (3):
- France (3):
  - CHU La Cavale Blanche, Brest
  - Centre Hospitalier Saint Jacques, Nantes
  - CHRU De Tours, Tours